CLINICAL TRIAL: NCT05693805
Title: Feasibility of Remote-Delivery Interventions: Tai Chi and Wellness for PTSD and Pain in Veterans
Brief Title: Feasibility of Remote Tai Chi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); VA Boston Healthcare System (U.S. Federal Agency); Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-42796; 1R34AT011547-01A1 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: PTSD; Pain, Chronic
Keywords: Tai Chi; PTSD; Chronic musculoskeletal pain; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain | interventions — Tai Ji; Health Promotion

STUDY DESIGN:
Intervention Model Description: Parallel Assignment for Phase One, Random Assignment for Phase Two.
Who Masked: Outcomes Assessor
Masking Description: The blinded evaluator will utilize remote videoconferencing to conduct structured interviews and assess each participant at baseline (prior to randomization), and post-treatment, and (for Phase Two only) at 3-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi Group (Experimental): Participants randomized to this arm will receive a standardized Tai Chi protocol developed for veterans, adapted by the investigators, and administered by experienced VA Tai Chi instructors.
  Interventions: Behavioral: Tai Chi
- Wellness Group (Active Comparator): Participants randomized to this arm will receive a wellness program that has been successfully used by the investigators in other studies of veterans with chronic pain.
  Interventions: Behavioral: Wellness program

INTERVENTIONS:
Behavioral: Tai Chi — The remote delivery Tai Chi protocol that will be developed in this study for Veterans with PTSD and pain will be adapted from a protocol that has been well-tested in previous trials All components of the program derive from the classical Yang-style Tai Chi 108 postures, which has been shown to be a moderate intensity exercise. Sessions will last 60 minutes, twice a week for 12 weeks. Experienced instructors will follow the Tai Chi protocol with rigorous quality control procedures. We will provide the patients with printed materials on the Tai Chi program, including Tai Chi principles, practice techniques, and safety precautions. Every session will include: warm up and a review of Tai Chi principles; breathing techniques; meditation with Tai Chi movement; and relaxation.
  Arms: Tai Chi Group
Behavioral: Wellness program — The Wellness intervention that will be developed for this study will consist of 60-minute sessions that meet twice a week for 12 weeks, and will be facilitated by doctoral level psychology staff and/or psychology trainees who will be supervised by staff. The Wellness intervention will be based on the VA Whole Health Program which helps individuals identify and achieve their personal health goals. The Whole Health Program include modules that address physical activity, personal development, healthy eating and drinking, stress management, relationships, personal surroundings, and spirituality. Using the SMART goals model, participants will set health and wellness goals each week. Discussions about ways to address potential barriers will be included in this condition.
  Arms: Wellness Group

SUMMARY:
In the proposed trial, the investigators plan to refine interventions, then conduct a small randomized trial to provide critical information to inform a future large-scale randomized efficacy trial of Tai Chi for Post Traumatic Stress Disorder (PTSD) and chronic pain. Building on the combined experience the proposed study will progress in new directions to:

1. Adapt, refine, and standardize two 12-week treatment protocols (Tai Chi and a Wellness control condition) for Veterans diagnosed with PTSD and chronic musculoskeletal pain during Phase One. Tai Chi and Wellness interventions will be adapted for delivery via a videoconferencing platform for the population and piloted in a 'dry run'.
2. Determine the feasibility and acceptability of a remotely delivered randomized trial of these two interventions and the assessment protocols during Phase Two.
3. Utilize information from this trial to plan and design a large randomized control study evaluating the efficacy of Tai Chi compared to Wellness for improving outcomes for Veterans with PTSD and chronic musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status as indicated by self-report
* PTSD Case Definition. Veterans who meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnostic criteria according to DSM-5 diagnostic algorithm for current PTSD as assessed on the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) will be eligible for the study. A diagnosis of current PTSD requires: a traumatic stressor (Criterion A) and the requisite number of symptoms at a severity level of 2 or higher in each symptom cluster. Each symptom is rated on a severity scale of 0 (no symptoms) to 4 (extreme), with 2 representing clinically significant and clearly present symptomatology. An individual must endorse at least one reexperiencing (Criterion B) symptom, at least one avoidance (Criterion C) symptom, at least two symptoms of negative alterations in cognition and mood (Criterion D), and at least two hyperarousal (Criterion E) symptoms. In addition, these symptoms must have been present for at least one month (Criterion F) and cause either clinically significant distress or functional impairment (Criterion G).
* Chronic pain as indicated by complaints of musculoskeletal pain in one or more body regions for six months or more.
* Willing to abstain from initiating evidence-based and mindfulness-based psychotherapy for PTSD, pain and related disorders until completion of the study (i.e., prolonged exposure, cognitive processing therapy, cognitive-behavioral treatment for insomnia or pain, acceptance and commitment therapy, dialectical behavior therapy, mindfulness-based stress reduction). Once enrolled, however, if other providers prescribe treatment or if participants require additional intervention (such as to manage a safety or substance abuse condition), treatment will be allowed, and appropriate referrals will be made. Individuals who are currently engaging in short-term (e.g., 12-week protocol) evidence-based treatment will not be eligible until treatment has ended.
* Access to internet and home computer or tablet device that will allow telehealth delivery of intervention.
* Available to attend either intervention group at the times they are scheduled.
* Enrolled and eligible to receive care in Veterans Health Administration (VHA). The investigators will facilitate enrollment for Veterans not currently enrolled but wish to take part in the study.

Exclusion Criteria:

* Lacks the capacity to provide consent.
* Diagnosed major medical disorder (e.g., neurological disorder, cancer, chronic infectious disease or liver disease) or has a moderate or severe traumatic brain injury, which could otherwise explain the health symptoms or interfere with their ability to safely engage in Tai Chi exercises.
* Change in psychotropic or pain medication during the past month. This will minimize amount of symptom change due to medication alterations. (Once enrolled, medication changes are nonetheless expected and will be monitored.)
* Regular current Tai Chi, formal mindfulness meditation program, or yoga practice, defined as at least three hours per week for more than three months. (Veterans with prior experience who do not currently engage in regular practice at this level will be eligible.)
* High risk from a mental health perspective e.g., recent psychiatric hospitalization, high risk flag or a note in their VA electronic health record indicating current high-risk factors, entered into a drug or alcohol detoxification or rehabilitation program, or attempted suicide within the previous year as indicated in their VA electronic health record.
* Pregnant or breastfeeding or plans to become pregnant within the year, assessed via self-report. Enrollment of pregnant or breastfeeding participants could potentially complicate outcomes, as new symptoms are likely to arise during the course of the intervention that are attributable to the pregnancy or breastfeeding and not the intervention or symptoms related to PTSD.
* Reports difficulty standing on feet for the majority of a Tai Chi class (approximately 60 minutes).
* Reports that they have been told by a doctor that they should not engage in physical activity unless recommended by a medical team.
* Reports other reason they cannot safely participate in physical activity.
* Concurrent participation in another clinical trial
* Participants who engage in behavior that is disrespectful or disrupts the group may be terminated from the study.
* Participants who demonstrate evidence of falsifying data may be terminated from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Niles, PhD, Principal Investigator — BUCA School of Medicine, Psychiatry; Boston Veterans Administration
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Veterans Health Administration (VHA) investigators interested in these data are invited to reach out to discuss data use agreements for the possibility of data sharing. Due to VHA rules related to data sharing and the sensitivity of health records data, data from this project cannot be shared on an open platform.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2027 to December 2028
Access Criteria: Investigators interested in these data are invited to reach out to discuss data use agreements for the possibility of data sharing.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tai Chi Group | Wellness Group
Started | 21 | 21
Completed | 16 | 19
Not Completed | 5 | 2
Not completed — Completed is defined as being engaged at the 3-month follow up.. | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai Chi Group | Wellness Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (14.3) | 58.1 (10.6) | 59.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 5 | 5
  White | 13 | 11 | 24
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Participant Satisfaction Post Treatment With Interventions Being Tested
Description: Assessed by the self-administered Client Satisfaction Questionnaire (CSQ), an 8-item scale with individual responses ranging from 1 to 4. Higher scores are associated with greater satisfaction with the treatment.
Time Frame: Post-treatment (about 12 weeks)
Population: CSQ data are not available for 3 participants in the Tai Chi Groups and 3 participants in the Wellness Group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Group | Wellness Group
Number analyzed (Participants) | 18 | 18
score on a scale | 3.61 (0.51) | 3.40 (0.56)

2. Primary Outcome: Percentage of Participants Satisfaction at Follow-up With Interventions Being Tested
Description: Percentage of participants that have a mean CSQ item-score of 3 or greater on the 1-4 scale of the 8 original items at post-treatment.
Time Frame: Post-treatment (about 12 weeks)
Population: CSQ data are not available for 3 participants in the Tai Chi Groups and 3 participants in the Wellness Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Tai Chi Group | Wellness Group
Number analyzed (Participants) | 18 | 18
Participants | 16 | 16

3. Primary Outcome: Number of Participants That Attended at Least 70% of the Treatment Sessions
Description: The number of participants that attended sessions was monitored by study staff.
Time Frame: Post-treatment (about 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Tai Chi Group | Wellness Group
Number analyzed (Participants) | 21 | 21
Participants | 14 | 15

4. Primary Outcome: The Percentage of Participants That Completed All Assessments
Description: Number of participants that completed all assessments (baseline through follow-up) was monitored by study staff.
Time Frame: Follow-up (about 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Tai Chi Group | Wellness Group
Number analyzed (Participants) | 21 | 21
Participants | 16 | 18

5. Secondary Outcome: Credibility of Treatment
Description: Credibility will be defined as a mean item-score of 6 or greater on the 1-9 scale of the 6 item Credibility/Expectancy Questionnaire (CEQ). Items 1-3 are specific to credibility and items 4-6 to expectancy.
Time Frame: 4 weeks
Population: CEQ data are not available for 2 participants in the Tai Chi Groups and 3 participants in the Wellness Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Tai Chi Group | Wellness Group
Number analyzed (Participants) | 19 | 18
Participants | 11 | 10

6. Secondary Outcome: Expectancy of Treatment
Description: Expectancy will be defined as a mean item-score of 6 or greater on the 1-9 scale of the 6 item Credibility/Expectancy Questionnaire (CEQ). Items 1-3 are specific to credibility and items 4-6 to expectancy.
Time Frame: 4 weeks
Population: CEQ data are not available for 2 participants in the Tai Chi Groups and 3 participants in the Wellness Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Tai Chi Group | Wellness Group
Number analyzed (Participants) | 19 | 18
Participants | 4 | 4

7. Secondary Outcome: Percentage of Participants Who Completed the Weekly Log Sheet
Description: Participants will complete the weekly log sheets that will be monitored by study staff. For the Tai Chi Group participants will record the number of minutes per day spent on home practice. For the Wellness Group, participants will record weekly goals.
Time Frame: Post treatment (about 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Tai Chi Group | Wellness Group
Number analyzed (Participants) | 21 | 21
Participants | 16 | 16

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Tai Chi Group | Wellness Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT05693805/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT05693805/ICF_000.pdf